CLINICAL TRIAL: NCT06521398
Title: Postpartum Care in the NICU (PeliCaN) Transitions
Acronym: PeliCaN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Heather Burris, Associate Professor of Pediatrics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 855528
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Stress Disorders, Post-Traumatic; Premature Birth; Postpartum Depression; Postpartum Anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Premature Birth; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doula Intervention (Experimental): Participants randomized to the intervention will be offered doula support including care coordination to mental and medical health services in the neonatal intensive care unit (NICU), with a warm handoff to a community doula to continue the support once infants leave the Hospital of the University of Pennsylvania (HUP) NICU.
  Interventions: Other: Doula Support
- Control (No Intervention): Participants randomized to usual care will get the same care they normally would with their own provider, outside of research enrollment, and receive a resource guide with information about the importance of postpartum follow-up care.

INTERVENTIONS:
Other: Doula Support — Doula support including care coordination to mental and medical health services in the NICU, with a warm handoff to a community doula to continue the support once infants leave the HUP NICU.
  Arms: Doula Intervention

SUMMARY:
This is a randomized controlled trial of a dyad-centered, doula support and healthcare coordination model of care in a large urban neonatal intensive care unit (NICU), which serves a high-risk, low-income, majority Black population. In addition to doula support and coordination of care in the NICU, there will be a warm handoff to a community doula to continue the support once infants leave the Hospital of the University of Pennsylvania (HUP) NICU.

ELIGIBILITY:
Inclusion Criteria:

* HUP postpartum patients who are at least 16 years old at the time their newborns' birth
* Infant born at HUP
* Preterm birth <34 weeks
* English language speaking

Exclusion Criteria:

* Unable to read or sign informed consent
* Parents of infants transferred into HUP NICU
* If the medical team believes that the infant may not live or be transferred to another hospital in upcoming weeks
* HUP postpartum patients who are less than 16 years of age at the time of their newborns' birth

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Difference in Post Traumatic Stress Disorder Scores at 6 months postpartum | 6 months
  This will measured by the PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The symptom severity score ranges from 0-80 with 80 being a worse score.
Number of participants who have attendance with a primary care provider by 6 months postpartum | 6 months
  This will be assessed using the electronic health record and via survey and medical record review of outsider records.

SECONDARY OUTCOMES:
Difference in Depression scores at 6 months postpartum | 6 months
  Edinburgh Postnatal Depression Scale, higher scores reflect higher risk of depression, ranges from 0-30. A score of 13 is indicative of high risk for depression.
Receipt of ACOG-recommended postpartum care by patient's designated provider | 12 weeks postpartum
  Comparison between two groups, this will be coded as a Yes or No variable

CONTACTS AND LOCATIONS:
Overall Officials: Heather Burris, MD MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States